CLINICAL TRIAL: NCT06713369
Title: A Phase I, Open-label Study to Assess the Absolute Bioavailability of Saruparib (AZD5305) and Absorption, Distribution, Metabolism, and Excretion (ADME) of [14C]-Saruparib ([14C]-AZD5305) in Patients With Advanced Solid Malignancies
Brief Title: AZD5305 hADME in Patients With Advanced Solid Malignancies
Acronym: AZD5305
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D9723C00004
Record Dates: First submitted 2024-07-30; First posted 2024-12-03 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced or Metastatic Solid Tumor
Keywords: hADME; saruparib; AZD5305; advanced solid tumour / tumor; neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — AZD5305

STUDY DESIGN:
Intervention Model Description: Approximately 8 patients will be enrolled, all will be assigned to the same treatment arm with no randomization or masking. All eligible patients will begin dosing in Part A, followed by a washout period, followed by Part B.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Treatment Arm - AZD5305 (Experimental): Part A will assess absolute bioavailability via oral administration of Saruparib (AZD5305) and IV [14C]-saruparib microtracer.
  Part B will assess ADME via IV [14C]-saruparib administration
  Interventions: Drug: Saruparib (AZD5305); Drug: [14C]-AZD5305 microtracer; Drug: [14C]-AZD5305 (therapeutic dose)

INTERVENTIONS:
Drug: Saruparib (AZD5305) — PARP-inhibitor
  Other Names: Saruparib
Drug: [14C]-AZD5305 microtracer — IV radiolabeled microtracer
  Other Names: IV [14C]-Saruparib microtracer
Drug: [14C]-AZD5305 (therapeutic dose) — IV radiolabeled PARP inhibitor
  Other Names: IV [14C]-Saruparib (therapeutic dose)

SUMMARY:
This Phase I, open-label study aims to study to absolute bioavailability of Saruparib (AZD5305) and the absorption, distribution, metabolism and excretion (ADME) of [14C]-Saruparib in patients with advanced solid malignancies.

This will be done on an inpatient basis in 2 parts (single-dose oral administration with radiolabeled microtracer in Part A, single-dose IV radiolabeled administration in Part B) during which samples will be obtained of plasma, urine, feces and vomitus (where applicable).

DETAILED DESCRIPTION:
This is an open-label, 2-part study in participants with advanced solid malignancies and will be conducted at multiple study sites.

Participants will be assessed for study eligibility prior to admission to the study site during a 28-day screening period. Participants will take part in both Parts A and B of the study.

Part A will assess the absolute bioavailability and evaluate the PK parameters of oral Saruparib and a radiolabelled IV microdose of [14C]-Saruparib

Participants will be admitted to the study site pre-dose of Part A and will remain resident at the study site for PK sampling and safety assessments.

A washout period will be observed between doses of Saruparib in Parts A and B.

Part B will assess the ADME of oral [14C]-Saruparib. Participants will be readmitted to the study site for Part B and will remain resident at the study site for excreta (urine, faeces, and any vomitus) collections, PK sampling, and safety assessments. Participants may be discharged from the study site prior to the last indicated day if both the following discharge criteria are met:

1. ≥ 90% mass balance recovery, and
2. < 1% of the total radioactive dose is recovered in combined excreta (urine and faeces) in 2 consecutive 24-hour periods.

Participants will return to the study site for a Follow-up Visit after the last dose of Saruparib which will include routine safety assessments. After the completion of Parts A and B, and following the Follow-up Visit, participants may be allowed further access to Saruparib.

Additional safety data collection will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age (or the legal age of consent in the jurisdiction in which the study is taking place), at the time of signing the ICF.
2. Histologically or cytologically documented, locally advanced or metastatic solid tumour, excluding lymphoma, for which standard therapy does not exist or has proven ineffective or intolerable.
3. ECOG performance status of 0 or 1 with no deterioration over the 2 weeks prior to dosing.
4. Predicted life expectancy ≥ 12 weeks.
5. Adequate organ and marrow function as defined in the protocol
6. Willingness and ability to comply with study and follow-up procedures.
7. Able and willing to stay in hospital for specified residential periods following administration of Saruparib/[14C]-Saruparib
8. Regular bowel movements
9. Body weight within normal range specified in protocol
10. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies Reproduction
11. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in the protocol

Exclusion Criteria:

1. Participants with a history of MDS/AML or with features suggestive of MDS/AML (as determined by prior diagnostic investigation). Specific screening for MDS/AML is not required.
2. Participants with any known predisposition to bleeding
3. Any history of persisting severe cytopenia due to any cause
4. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of Saruparib.
5. History of another primary malignancy, with some exceptions
6. Persistent toxicities (CTCAE Grade ≥ 2), excluding alopecia, caused by previous anticancer therapy.
7. Spinal cord compression or brain metastases for at least 4 weeks prior to start of study intervention unless asymptomatic and stable
8. Abnormal cardiac function exclusions or cardiovascular disease
9. History of arrhythmia
10. Active HBV (positive HBsAg result) or HCV.
11. Evidence of active and uncontrolled HIV infection.
12. Active tuberculosis infection
13. Major surgical procedure (excluding placement of vascular access) or significant traumatic injury within 4 weeks of the first dose of study intervention or an anticipated need for major surgery during the study.
14. As judged by the investigator, any other evidence of diseases (such as severe or uncontrolled systemic diseases or active uncontrolled infections which, in the investigator's opinion, makes it undesirable for the participant to participate in the study or would jeopardise compliance with the protocol.
15. Any prior treatment with a PARP inhibitor or platinum chemotherapy.
16. Other anticancer therapy (chemotherapy, immunotherapy, hormonal anticancer therapy, radiotherapy [except for palliative local radiotherapy]), biological therapy or other novel agent is not permitted until the last PK sampling is completed.
17. Palliative radiotherapy with a limited field of radiation within 2 weeks or with wide field of radiation or to more than 30% of the bone marrow within 4 weeks before the first dose of study intervention
18. Concomitant use of medications or herbal supplements known to be CYP3A4 strong and moderate inhibitors or inducers
19. Concomitant use of drugs that are known to prolong or shorten QT and have a known risk of Torsades de Pointes
20. Participants who have participated in another absorption, distribution, metabolism, and excretion study within 1 year prior to screening.
21. Participation in another clinical study with a study intervention administered in the last 3 months or 5 half-lives prior to dosing, whichever is longer.
22. Participants with a known hypersensitivity to Saruparib or any of the excipients of the product.
23. Participants who have been administered any amount of a [14C]-labelled compound within the last 12 months.
24. Use of tobacco- or nicotine-containing products or alcohol may be exclusionary
25. Poor peripheral venous access (venous access via a port will be permitted).
26. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
27. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
28. Previous enrolment in the present study.
29. For female participants only: currently pregnant (confirmed with positive pregnancy test) or planning to become pregnant, breast-feeding, or intending to donate/retrieve ova before 6 months after the last dose of Saruparib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-10-02 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Absolute bioavailability (F) of Saruparib | Day 4
  Absolute bioavailability (F) of Saruparib
Total radioactivity recovery in urine and faeces | Day 8
  Total radioactivity recovery in urine and faeces
Pharmacokinetics of Saruparib(Part B) | Day 8
  AUCinf
PK parameters characterized by AUCinf | Day 4
  AUCinf
Ratio of AUCinf of plasma Saruparib relative to AUCinf of metabolite | Day 4
  Ratio of AUCinf of plasma Saruparib relative to AUCinf of metabolite
Mass balance parameters as characterized by amount excreted and cumulative amount excreted in urine, faeces and total (urine and faeces combined) | Day 8
  Cumulative amount excreted in urine, faeces and total (urine and faeces combined)
Amount excreted and cumulative amount excreted in urine, faeces and total (urine and faeces combined) expressed as a percentage of the administered dose | Day 8
  Amount excreted and cumulative amount excreted in urine, faeces and total (urine and faeces combined) expressed as a percentage of the administered dose.
Pharmacokinetics of Saruparib(Part B) | Day 8
  AUClast
Pharmacokinetics of Saruparib(Part B) | Day 8
  Cmax
Pharmacokinetics of Saruparib(Part B) | Day 8
  tmax
Pharmacokinetics of Saruparib(Part B) | Day 8
  t1/2(lambda)z
Pharmacokinetics of Saruparib(Part B) | Day 8
  Ratio of AUCinf of plasma Saruparib relative to AUCinf of plasma total radioactivity
Pharmacokinetics of Saruparib(Part B) | Day 8
  Ratio of AUCinf of whole blood total radioactivity relative to AUCinf of plasma total radioactivity
PK parameters characterized by AUClast | Day 4
  AUClast
PK parameters characterized by Cmax | Day 4
  Cmax
PK parameters characterized by tmax | Day 4
  tmax
PK parameters characterized by t1/2(lambda)z | Day 4
  t1/2(lambda)z

SECONDARY OUTCOMES:
Metabolic profiling of a single oral dose of [14C]-Saruparib (Part B) | Day 8
  Determining mass balance parameters following oral administration of a therapeutic dose containing 20uCi of 14C-AZD5305 followed by metabolite profiling and identification in plasma, urine, and feces to quantify the 14C-AZD5305 related material in each matrix to satisfy MIST considerations.
Characterize the safety of Saruparib in participants with advanced solid malignancies by incidence and severity of AEs, laboratory abnormalities, 12-lead ECG abnormalities, vital signs abnormalities, physical examination findings | Day 14
  incidence and severity of AEs, -incidence of laboratory abnormalities (based on hematology, clinical chemistry, and urinalysis test results), -12-lead ECG abnormalities, vital signs abnormalities, physical examination findings

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Research Site, Liverpool
  - Research Site, Manchester